CLINICAL TRIAL: NCT00471744
Title: HEAD-TO-HEAD Evaluation of the Antiepileptic Drugs Levetiracetam (LEV) vs. Sulthiame (STM) in a German Multi-Centre, Doubleblind Controlled Trial in Children With Benign Epilepsy With Centro-Temporal Spikes
Brief Title: HEAD-Study Optimizing the Treatment of Children With BECTS
Acronym: HEAD
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: low patient number after 2 years recruiting
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2005-004468-22; ISRCTN 97864911
Record Dates: First submitted 2007-05-08; First posted 2007-05-10 (Estimated); Last update posted 2009-01-29 (Estimated); Status verified 2009-01

CONDITIONS: Epilepsy, Rolandic
Keywords: benign epilepsy; pediatrics; children; rolandic epilepsy; levetiracetam; sulthiame
MeSH Terms: conditions — Epilepsy, Rolandic | interventions — Therapeutics; Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Treatment with levetiracetam or sulthiame over a six-month period.

SUMMARY:
The investigators hypothesize that Levetiracetam is as effective as Sulthiame in the treatment of children with BECTS. Patients entering the HEAD-Studie are either treated with Leveitracetam or Sulthiame over a 6 months period. Patients are equally randomised to one of the two treatment regimens. Administration of medication as blinded capsules.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 6 and 12 years
2. Weight between 15 kg and 60 kg
3. At least two preceding seizures within the last six months before study start
4. Typical electroencephalogram (EEG) with Rolando focus (centrotemporal spike or sharp-wave-focus)
5. Diagnosis of BECTS
6. Written informed consent from parents and child

Exclusion Criteria:

1. Other forms of epilepsy (e.g. continuous spikes and waves during slow sleep [CSWS], Landau-Kleffner-syndrome)
2. Preceding treatment with antiepileptic drugs
3. Mental Retardation (intelligence quotient [IQ] <85)
4. Focal neurological deficit
5. Relevant major internistic disease (e.g. hepatopathy, nephropathy, endocrinopathy)
6. Participation in another clinical trial within the last 30 days

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2006-06; Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of levetiracetam in the treatment of children with BECTS compared to sulthiame | 6 months

SECONDARY OUTCOMES:
Safety and tolerability | 6 months
Cognitive effects | 6 months
Efficacy on EEG pattern | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: F Heinen, Prof., Principal Investigator — Ludwigs-Maximilians-Universität München
Locations (1):
- Dr. von Haunersches Kinderspital, München, Germany

REFERENCES:
- [Derived] Milburn-McNulty P, Panebianco M, Marson AG. Sulthiame monotherapy for epilepsy. Cochrane Database Syst Rev. 2021 Sep 23;9(9):CD010062. doi: 10.1002/14651858.CD010062.pub3. PMID 34554571